CLINICAL TRIAL: NCT04511026
Title: Concurrent Use of Lymphoseek and Indocyanine Green for Sentinel Lymph Node Detection in Endometrial Cancer - a Prospective Study
Brief Title: Concurrent Use Lymphoseek & Indocyanine Green in Sentinel Lymph Node Detection in Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Efficacy
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Amer Karam, Clinical Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-53978; GYNEND0006 (Other: OnCore); IRB-53978 (Other: Stanford IRB)
Record Dates: First submitted 2020-08-07; First posted 2020-08-12 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — technetium-diethylenetriaminepentaacetic acid-mannosyl-dextran; Tomography, Emission-Computed, Single-Photon; Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Lymphoseek/SPECT-CT/Indocyanine (Experimental): The subject will receive f 0.5 mL each Lymphoseek into the uterine cervix prior to surgery and subsequent SPECT/CT imaging preoperatively. Intraoperatively, following anesthesia induction, Indocyanine Green (0.5 mL) will be injected into the uterine cervix. Using near-infrared imaging, efferent lymphatic vessels and lymph nodes will be visualized and confirmed by detected radioactivity using a laparoscopic gamma counter. The preoperatively obtained SPECT/CT images will help guide the surgery.
  Interventions: Drug: Lymphoseek; Device: Single Photon Emission Computed Tomography (SPECT); Drug: Indocyanine Green (ICG); Device: Neoprobe Gamma Detection System NPB11L(Model1102)

INTERVENTIONS:
Drug: Lymphoseek — Radioactive diagnostic agent
  Other Names: technetium Tc 99m tilmanocept
Device: Single Photon Emission Computed Tomography (SPECT) — Imaging test
Drug: Indocyanine Green (ICG) — Cyanine dye used in medical diagnostics manufactured by Akorn Inc.
Device: Neoprobe Gamma Detection System NPB11L(Model1102) — Neoprobe Gamma Detection System NPB11L(Model1102) made by Devicor Medical Products, Inc.
  Other Names: Laparoscopic handheld gamma counter

SUMMARY:
The goal of this study is to (i) improve detection of sentinel nodes and (ii) reduce additional surgical dissection that is needed in case a sentinel lymph node cannot be detected.

DETAILED DESCRIPTION:
Primary Objective: To determine the detection rate of bilateral sentinel lymph nodes with the concurrent use of Lymphoseek and Indocyanine Green.

Secondary Objective: (1) To determine the overall detection rate of sentinel lymph nodes with concurrent use of Lymphoseek and Indocyanine Green (2) To determine location and number of Lymphoseek-positive sentinel lymph nodes preoperatively by single-photon emission computed tomography (SPECT/CT imaging) and intraoperatively by a laparoscopic handheld gamma detection device and near- infrared fluorescent imaging (3) To determine the concordance of Lymphoseek-positive sentinel lymph nodes with intraoperatively detected Indocyanine Green-positive sentinel lymph nodes.

ELIGIBILITY:
Inclusion Criteria:

* The patient has histological diagnosis of cancer of the endometrium of any histology or grade.
* The patient should have received no prior treatment for her endometrial cancer.
* The patient has clinically uterine confined disease.
* The patient is a candidate for minimal invasive surgery, with sentinel lymph node assessment with IC-GREEN planned as part of standard of care.
* The patient has an Eastern Cooperative Group (ECOG) performance status of 0-2.
* If age less than or equal to 55 years, the patient has a negative pregnancy test within 72 hours before administration of Lymphoseek, has been surgically sterilized, or has been postmenopausal for at least 1 year.
* The patient has provided written informed consent.
* The patient is at least 18 years of age at the time of consent

Exclusion Criteria:

* The patient has clinical or radiological evidence of metastatic disease.
* The patient has a history of a prior loop electrosurgical excision procedure (LEEP) or cone procedure performed on her cervix.
* The patient has participated in another investigational drug study within 30 days of scheduled surgery.
* The patient has an iodine allergy.
* The patient is pregnant or lactating.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2021-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amer K Karam, MD, Principal Investigator — Stanford Universiy
Locations (1):
- Stanford University, School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Reddy RA, Moon AS, Chow S, Heilbroner L, Howitt B, Diver E, Dorigo O, Litkouhi B, Renz M, Karam A. Technetium Tc 99m tilmanocept fails to detect sentinel lymph nodes in endometrial cancer. Gynecol Oncol Rep. 2022 Jul 30;43:101054. doi: 10.1016/j.gore.2022.101054. eCollection 2022 Oct. PMID 35958955

RESULTS

PARTICIPANT FLOW:
Groups:
- Lymphoseek/SPECT-CT/Indocyanine: Participants received f 0.5 mL each Lymphoseek into the uterine cervix prior to surgery and subsequent SPECT/CT imaging preoperatively. Intraoperatively, following anesthesia induction, Indocyanine Green (0.5 mL) was injected into the uterine cervix. Using near-infrared imaging, efferent lymphatic vessels and lymph nodes were visualized and confirmed by detected radioactivity using a laparoscopic gamma counter. The preoperatively obtained SPECT/CT images helped guide the surgery.
Period: Overall Study
Arm/Group | Lymphoseek/SPECT-CT/Indocyanine
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lymphoseek/SPECT-CT/Indocyanine
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Histology [Count of Participants; unit: Participants] — Low-grade endometrioid carcinomas (EECs) grade is based on the proportion of solid areas: low grade = grade 1 (≤5%) and grade 2 (6%-50%); and high grade = grade 3 (>50%).
  Participants
    Endometrioid Grade 1 | 3
    Endometrioid Grade 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bilateral SLNs
Description: A sentinel lymph node will be defined as being detected if it is detected on the pre-operative SPECT/CT imaging scan or intraoperatively using near-infrared imaging or the handheld gamma detection device.
Time Frame: during surgery, an average of 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphoseek/SPECT-CT/Indocyanine
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: Overall Detection of SLN Detection
Description: For each subject, an assessment will be made of whether there was overall sentinel node detection. A sentinel lymph node will be defined as being detected if it is detected on the pre-operative SPECT/CT imaging scan or intraoperatively using near-infrared imaging or the handheld gamma detection device. If at least one SLN is detected (on any side), then this outcome will be considered a 'Yes'.
Time Frame: during surgery, an average of 3 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Lymphoseek/SPECT-CT/Indocyanine
Number analyzed (Participants) | 6
Participants | 6

3. Secondary Outcome: Number of SLNs Detected by Lymphoseek:
Description: The number of sentinel lymph nodes detected by Lymphoseek will be assessed. A sentinel lymph node will be defined as being detected by Lymphoseek if it is detected using the pre-operative SPECT/CT imaging scan and/or intraoperatively using the gamma detection device.
Time Frame: during surgery, an average of 3 hours
Measure: Number; unit: SLNs
Arm/Group | Lymphoseek/SPECT-CT/Indocyanine
Number analyzed (Participants) | 6
SLNs | 0

4. Secondary Outcome: Location of SLNs Detected by Lymphoseek:
Description: The location and number of sentinel lymph nodes detected by Lymphoseek will be assessed. A sentinel lymph node will be defined as being detected by Lymphoseek if it is detected using the pre-operative SPECT/CT imaging scan and/or intraoperatively using the gamma detection device.
Time Frame: during surgery, an average of 3 hours
Population: Data are not available as no SLNs were detected using Lymphseek
Arm/Group | Lymphoseek/SPECT-CT/Indocyanine
Number analyzed (Participants) | 0

5. Secondary Outcome: Number of SLNs Detected by Indocyanine Green
Description: Number of SLNs detected by Indocyanine Green: The location and number of sentinel lymph nodes detected by Indocyanine Green will be assessed. A sentinel lymph node will be defined as being detected by Indocyanine Green if it is detected intraoperatively using near-infrared imaging only and not by the gamma detection device.
Time Frame: during surgery, an average of 3 hours
Measure: Number; unit: SLNs
Arm/Group | Lymphoseek/SPECT-CT/Indocyanine
Number analyzed (Participants) | 6
SLNs | 28

6. Secondary Outcome: Location of SLNs Detected by Indocyanine Green
Description: Location of SLNs detected by Indocyanine Green: The location and number of sentinel lymph nodes detected by Indocyanine Green will be assessed. A sentinel lymph node will be defined as being detected by Indocyanine Green if it is detected intraoperatively using near-infrared imaging only and not by the gamma detection device.
Time Frame: during surgery, an average of 3 hours
Measure: Count of Units; unit: SLNs
Units Other Than Participants: SLNs
Groups:
- Right-Sided SLN Locations; Left-Sided SLN Locations: Participants received f 0.5 mL each Lymphoseek into the uterine cervix prior to surgery and subsequent SPECT/CT imaging preoperatively. Intraoperatively, following anesthesia induction, Indocyanine Green (0.5 mL) was injected into the uterine cervix. Using near-infrared imaging, efferent lymphatic vessels and lymph nodes were visualized and confirmed by detected radioactivity using a laparoscopic gamma counter. The preoperatively obtained SPECT/CT images helped guide the surgery.
Arm/Group | Right-Sided SLN Locations | Left-Sided SLN Locations
Number analyzed (Participants) | 6 | 6
Number analyzed (SLNs) | 11 | 17
SLNs
  Common Iliac | 2 | 1
  External Iliac | 8 | 9
  Hypogastric | 0 | 1
  Obturator | 1 | 6

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Lymphoseek/SPECT-CT/Indocyanine
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
This study did not meet its planned enrollment and did not achieve statistical power.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/26/NCT04511026/Prot_SAP_000.pdf